CLINICAL TRIAL: NCT01168037
Title: Medical and Economical Evaluation of Endovascular Therapy of Complex Aortic Aneurysms (Para- & Supra- Renal Abdominal Aortic Aneurysms, Type 4 THORACO-Abdominal Aneurysms) by Fenestrated & Branched Stent-grafts
Brief Title: Medical & Economical Evaluation of Fenestrated & Branched Stent-grafts to Treat Complex Aortic Aneurysms
Acronym: Windows1
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: IC090126
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Aortic Aneurysms
Keywords: Aorta; Aneurysm; endovascular; stent-graft
MeSH Terms: conditions — Aortic Aneurysm; Aneurysm | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Open repair: Open Surgical Repair (aortic replacement with revascularization of visceral arteries)
  Interventions: Procedure: Open Surgical Repair
- Endovascular (Windows 1): Endovascular therapy branched or fenestrated stent-graft
  Interventions: Device: Endovascular aortic repair with branched/fenestrated stent-graft
- Endovascular (Windows 3): Endovascular therapy branched or fenestrated stent-graft (vascutek anaconda)
  Interventions: Device: Endovascular aortic repair with branched/fenestrated stent-graft

INTERVENTIONS:
Device: Endovascular aortic repair with branched/fenestrated stent-graft — Insertion via bilateral femoral access, stent-graft deployment under fluoroscopic guidance, complementary stenting of visceral arteries, control angiogram
  Other Names: Endovascular aortic repair
  Groups: Endovascular (Windows 1); Endovascular (Windows 3)
Procedure: Open Surgical Repair — aortic replacement with revascularization of visceral arteries
  Groups: Open repair

SUMMARY:
The aim of this study is to prospectively compare the perioperative mortality severe morbidity and the costs of endovascular versus conventional surgical repair of pararenal, supra-renal and type 4 THORACO-abdominal aortic aneurysms.

The primary goal of the study is to demonstrate a significant drop in 30-day mortality and life threatening morbidity in the endovascular arm of the study. Our hypothesis, derived from the literature, that the average 30-days mortality is 3% after endovascular repair and 10% after open surgery justifies the design of a prospective study between endovascular therapy (250 patients (amendment) treated in 8 University hospitals with significant experience of the technique) and open repair (660 similar patients analyzed form the national database of the MOH).

DETAILED DESCRIPTION:
The aim of this study is to prospectively compare the perioperative mortality severe morbidity and the costs of endovascular versus conventional surgical repair of pararenal, supra-renal and type 4 THORACO-abdominal aortic aneurysms.

The primary goal of the study is to demonstrate a significant drop in 30-day mortality and life threatening morbidity in the endovascular arm of the study. Our hypothesis, derived from the literature, that the average 30-days mortality is 3% after endovascular repair and 10% after open surgery justifies the design of a prospective study between endovascular therapy (250 patients (amendment) treated in 8 University hospitals with significant experience of the technique) and open repair (660 similar patients analyzed form the national database of the MOH).

In-hospital morbidity are similarly expected to be lower in the endovascular group. We also wish to demonstrate that endovascular repair does not represent a significant over-cost, as compared to open repair. The cost of the implantable medical device (IMD), of follow-up screening, and of eventual repeated interventions should be compensated by a reduced stay in intensive care unit ICU, and by a reduced in-hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

The following anatomical inclusion criteria must be met:

* Absence of significant angulations (< 60°) of aorta or of iliac arteries
* Absence of tight stenosis (>70%) of more than one target artery (renal or visceral artery to be perfused from the side holes of the stent-graft)
* Diameter of target arteries over 5 mm
* Iliac and femoral arteries allowing insertion of the delivery system (> 7 mm) or suitable for insertion of an access conduit

Exclusion Criteria:

* Limited expected life expectancy
* Emergency cases
* Refuse to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with an Abdominal aortic aneurysm over 5 cm in diameter or with a diameter increase over 1 cm in 1 year and a PSRAA defined by:
  * Infrarenal aortic neck < 15 mm
  * or extent of the aneurismal process to the suprarenal aorta
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2009-06-17 (Actual); Primary Completion 2015-02-09 (Actual); Study Completion 2015-02-09 (Actual)

PRIMARY OUTCOMES:
30-day postoperative mortality | 30-day postoperative

SECONDARY OUTCOMES:
complications | 30-day postoperative
Length of Intensive Care Unit (ICU) stay | 30-day postoperative
Length of Hospital stay | 30-day postoperative
Overall cost | 30-day postoperative
Reinterventions | 2-year follow up
Global survival | 2-year follow up
Mortality in touch with aneurysm | 2-year follow up
Annual cost (1 month, 6 month, 1 year and 2 year Follow-up screening ) | 2-year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Becquemin, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] O'Neill S, Greenberg RK, Haddad F, Resch T, Sereika J, Katz E. A prospective analysis of fenestrated endovascular grafting: intermediate-term outcomes. Eur J Vasc Endovasc Surg. 2006 Aug;32(2):115-23. doi: 10.1016/j.ejvs.2006.01.015. Epub 2006 Mar 31. PMID 16580236
- [Derived] Michel M, Becquemin JP, Clement MC, Marzelle J, Quelen C, Durand-Zaleski I; WINDOW Trial Participants. Editor's choice - thirty day outcomes and costs of fenestrated and branched stent grafts versus open repair for complex aortic aneurysms. Eur J Vasc Endovasc Surg. 2015 Aug;50(2):189-96. doi: 10.1016/j.ejvs.2015.04.012. Epub 2015 Jun 19. PMID 26100447
- [Derived] Marzelle J, Presles E, Becquemin JP; WINDOWS trial participants. Results and factors affecting early outcome of fenestrated and/or branched stent grafts for aortic aneurysms: a multicenter prospective study. Ann Surg. 2015 Jan;261(1):197-206. doi: 10.1097/SLA.0000000000000612. PMID 24670864
- [Derived] Banno H, Kobeiter H, Brossier J, Marzelle J, Presles E, Becquemin JP. Inter-observer variability in sizing fenestrated and/or branched aortic stent-grafts. Eur J Vasc Endovasc Surg. 2014 Jan;47(1):45-52. doi: 10.1016/j.ejvs.2013.10.008. Epub 2013 Oct 23. PMID 24268517